CLINICAL TRIAL: NCT01814683
Title: Improving the Radical Cure of Vivax Malaria: A Multicentre Randomised Comparison of Short and Long Course Primaquine Regimens
Brief Title: IMPROV (Improving the Radical Cure of Vivax Malaria)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Menzies School of Health Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BAKMAL 1301
Record Dates: First submitted 2013-03-18; First posted 2013-03-20 (Estimated); Last update posted 2019-09-17 (Actual); Status verified 2018-07

CONDITIONS: Uncomplicated Vivax Malaria
Keywords: Vivax malaria; Primaquine; Placebo; Recurrence
MeSH Terms: conditions — Malaria, Vivax; Recurrence | interventions — Primaquine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Primaquine 7 day (Experimental): Standard blood schizontocidal therapy plus 7 days of supervised primaquine (7mg/kg total dose) administered once per day (1.0 mg/kg OD) followed by 7 days of placebo.
  Interventions: Drug: Primaquine
- Placebo controlled arm (Placebo Comparator): Standard blood schizontocidal therapy plus 14 days placebo.
  Interventions: Drug: Placebo
- Primaquine 14 day (Active Comparator): Standard blood schizontocidal therapy plus 14 days of supervised primaquine (7mg/kg total dose) administered once per day (0.5 mg/kg).
  Interventions: Drug: Primaquine

INTERVENTIONS:
Drug: Primaquine — 14 days of supervised primaquine (7mg/kg total dose) administered once per day (0.5 mg/kg).
  Arms: Primaquine 14 day
Drug: Primaquine — 7 days of supervised primaquine (7mg/kg total dose) administered once per day (1.0 mg/kg OD) followed by 7 days of placebo.
  Arms: Primaquine 7 day
Drug: Placebo — 14 days placebo.
  Arms: Placebo controlled arm

SUMMARY:
The main determinant of primaquine efficacy is the total dose of primaquine administered, rather than the dosing schedule. Previous trials have demonstrated that the standard low dose regimen of primaquine (3.5 mg/kg total) fails to prevent relapses in many different endemic locations. For this reason the 2010 WHO antimalarial guidelines now recommend a high dose regimen of 7 mg/kg (equivalent to an adult dose of 30mg per day), although many countries still recommend lower doses for fear of causing more serious harm to unscreened G6PDd patients.

Shorter courses of higher daily doses of primaquine have the potential to improve adherence and thus effectiveness without compromising efficacy. Primaquine also has relatively weak but clinically relevant asexual stage activity against P. vivax so larger daily doses may substantially augment chloroquine's blood stage activity at low levels of resistance. In Thailand directly observed primaquine (1mg/kg/day) administered over 7 days was well tolerated and reduced relapses by day 28 to 4%. This is encouraging but not definitive since many relapses present after one month. Longer follow-up is needed to distinguish whether relapse was prevented or deferred. If the efficacy, tolerability and safety of short-course, high-dose primaquine regimens can be assured across the range of endemic settings, along with reliable point-of-care G6PDd diagnostics, then this new primaquine regimen would be a major advance in malaria treatment improving adherence to and thus the effectiveness of anti-relapse therapy.

Due to the long duration of standard primaquine treatment regimens, courses are difficult to supervise, are poorly adhered to and lack effectiveness. This proposed multicentre randomised clinical trial will provide evidence across a variety of endemic settings on the safety and efficacy of high dose-short course primaquine in G6PD normal patients. In a parallel single arm study the investigators will also gather safety data on the use of weekly primaquine in patients with G6PDd. This study aims to generate evidence that will directly inform global public health policy for the radical cure of P. vivax. A better understanding of the risks and benefits of primaquine is crucial in persuading policy makers and clinicians of the importance of the radical cure of vivax malaria that will reduce the parasite reservoir and decrease transmission.

The funder is Medical Research Council, UK. Grant number: MRC Reference: MR/K007424/1

DETAILED DESCRIPTION:
Plasmodium vivax malaria is a major cause of morbidity and now recognised as an important contributor to mortality in endemic areas. Unlike P. falciparum malaria, P. vivax infections form dormant liver stages (hypnozoites) which cause relapses of the infection weeks to months after the initial attack for up to about 2 years. Relapse rates in South-East Asia commonly exceed 50%, often making relapse the main cause of vivax illness. Repeated relapse is particularly damaging to the health and development of children in vivax endemic areas. The first line treatment of vivax malaria is a combination of chloroquine (providing blood schizontocidal activity), and primaquine (providing liver hypnozoitocidal activity). However chloroquine resistance is increasing in many vivax endemic areas and adherence to 14 day primaquine regimens is very poor. This is a major threat to current malaria control and elimination initiatives. Primaquine, an 8 aminoquinoline, is currently the only licensed drug with activity against hypnozoites. An important constraint on the global deployment of primaquine is its potential to cause haemolysis in patients with glucose-6-phosphate dehydrogenase deficiency (G6PDd), which typically occurs in 2-15% (and up to 40%) of patients in endemic zones. Individuals who have less than 10% of normal enzyme activity are at risk of life-threatening haemolysis whereas those with milder variants may have negligible effects. In practice the lack of available robust diagnostics for G6PDd, concerns over drug toxicity, and the misperceived benign nature of P. vivax infection results in healthcare providers rarely prescribing primaquine even when recommended in policy.

The main determinant of primaquine efficacy is the total dose of primaquine administered, rather than the dosing schedule. Previous trials have demonstrated that the standard low dose regimen of primaquine (3.5 mg/kg total) fails to prevent relapses in many different endemic locations. For this reason the 2010 WHO antimalarial guidelines now recommend a high dose regimen of 7 mg/kg (equivalent to an adult dose of 30mg per day), although many countries still recommend lower doses for fear of causing more serious harm to unscreened G6PDd patients.

Shorter courses of higher daily doses of primaquine have the potential to improve adherence and thus effectiveness without compromising efficacy. Primaquine also has relatively weak but clinically relevant asexual stage activity against P. vivax so larger daily doses may substantially augment chloroquine's blood stage activity at low levels of resistance. In Thailand directly observed primaquine (1mg/kg/day) administered over 7 days was well tolerated and reduced relapses by day 28 to 4%. This is encouraging but not definitive since many relapses present after one month. Longer follow-up is needed to distinguish whether relapse was prevented or deferred. If the efficacy, tolerability and safety of short-course, high-dose primaquine regimens can be assured across the range of endemic settings, along with reliable point-of-care G6PDd diagnostics, then this new primaquine regimen would be a major advance in malaria treatment improving adherence to and thus the effectiveness of anti-relapse therapy.

The radical cure of P. vivax in patients with known G6PDd is challenging. Current WHO guidelines recommend a weekly dose of 0.75 mg/kg for 8 weeks which mitigates primaquine-induced haemolysis whilst retaining efficacy. The weekly dosing schedule was derived from studies in the USA in a small number of healthy adults with the mildly primaquine-sensitive African A- G6PDd variant. Since host vulnerability to haemolysis varies between the over 100 different G6PDd variants, the available evidence is inadequate to ensure the universal safety of a 0.75mg/kg dose either as a single dose, as advocated for reducing the transmission of falciparum malaria, or a weekly dose for the radical cure of vivax malaria.

Due to the long duration of standard primaquine treatment regimens, courses are difficult to supervise, are poorly adhered to and lack effectiveness. This proposed multicentre randomised clinical trial will provide evidence across a variety of endemic settings on the safety and efficacy of high dose-short course primaquine in G6PD normal patients. In a parallel single arm study the investigators will also gather safety data on the use of weekly primaquine in patients with G6PDd. This study aims to generate evidence that will directly inform global public health policy for the radical cure of P. vivax. A better understanding of the risks and benefits of primaquine is crucial in persuading policy makers and clinicians of the importance of the radical cure of vivax malaria that will reduce the parasite reservoir and decrease transmission.

RESULTS:

The incidence rate of symptomatic recurrent P. vivax malaria was 0.18 (95% CI, 0.15 to 0.21) episodes PPY following PQ7, 0.16 (95% CI, 0.13 to 0.18) PPY following PQ14 and 0.96 (95% CI, 0.83 to 1.08) PPY in the control arm

The incidence rate of both symptomatic and asymptomatic recurrent vivax malaria at 1 year was 0.23 (95%CI, 0.19 to 0.27) episodes PPY following PQ7 and 0.19 (95% CI: 0.16 to 0.23) episodes PPY following PQ14 (p=0.208)

In the time to first event analysis, the cumulative risk of symptomatic P. vivax at 1 year was 14.28% (95%CI, 11.75 to 17.29) after PQ7 and 12.72% (95%CI, 10.19 to 15.82) after PQ14 (p=0.197), both significantly lower than 48.73% (95%CI, 43.40 to 54.36) in the control arm (HR=0.18 [95%CI, 0.13 to 0.26; p<0.001] and HR=0.14 [95%CI, 0.09 to 0.22; p<0.001], respectively)

There were 27 SAEs: 18 (1.9%) in the PQ7 arm, 5 (0.5%) in the PQ14 arm and 4 (0.9%) in the control arm. Ten of these SAEs occurred within 42 days and were considered study drug related: 1.0% (9/935, PQ7), 0.1% (1/937, PQ14) (p=0.001) and none (0/464) in the control arm.

ELIGIBILITY:
Inclusion Criteria:

* Participant (or parent/guardian of children below age of consent) is willing and able to give written informed consent to participate in the trial; verbal consent in the presence of a literate witness is required for illiterate patients. In addition, written assent (or verbal assent in the presence of a literate witness for illiterates) from children 12 to 17 years as per local practice.
* Monoinfection with P. vivax of any parasitaemia in countries which use Chloroquine (CQ) as blood schizontocidal therapy. Mixed infections with P. vivax and P. falciparum can be enrolled in countries which use an artemisinin combination therapy.
* Diagnosis based on rapid diagnostic tests.
* Over 6 months of age.
* Weight 5 kg or greater.
* Fever (axillary temperature 37.5 degrees C) or history of fever in the last 48 hours.
* Able, in the investigators opinion, and willing to comply with the study requirements and follow-up.

Exclusion Criteria:

* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Inability to tolerate oral treatment.
* Previous episode of haemolysis or severe haemoglobinuria following primaquine
* Signs/symptoms indicative of severe/complicated malaria or warning signs requiring parenteral treatment- Haemoglobin concentration less than 9 g/dL
* Known hypersensitivity or allergy to the study drugs
* Blood transfusion in last 90 days, since this can mask G6PD deficient status
* A febrile condition due to diseases other than malaria (e.g. measles, acute lower respiratory tract infection, severe diarrhoea with dehydration)
* Presence of any condition which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal or hepatic disease; severe malnutrition; HIV/AIDS; or severe febrile condition other than malaria); coadministration of other medication known to cause haemolysis or that could interfere with the assessment of antimalarial regimens.
* Currently taking medication known to interfere significantly with the pharmacokinetics of primaquine and the schizontocidal study drugs.
* Prior antimalarial medications in the previous 7 days.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2388 (Actual)
Dates: Start 2014-07 (Actual); Primary Completion 2018-02-28 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Incidence rate (per person-year) of symptomatic recurrent P. vivax | 12 months
  The incidence rate (i.e. per person-year) of symptomatic recurrent P. vivax parasitaemia (detected by microscopy) over 12 months of follow-up in the 7 versus 14-day primaquine groups for all sites combined and stratified by site.

SECONDARY OUTCOMES:
The incidence rate (per person-year) of any recurrent P. vivax malaria. | 12 months
  The incidence rate (per person-year) of any recurrent (i.e. symptomatic and asymptomatic) P. vivax parasitaemia over 12 months of follow-up in the 7 and 14-day primaquine regimens for all sites combined and stratified by site.
Incidence risk of any recurrent symptomatic of P. vivax malaria compared to control arm | 12 months
  The incidence rate (per person-year) of any recurrent symptomatic P. vivax parasitaemia over 12 months of follow-up in either the 7 or the 14-day primaquine regimens compared with the control arm, for all sites combined and stratified by site.
The Haematological recovery in patients with vivax malaria | 12 months
  Haematological recovery will be assessed as the incidence risk of severe anaemia (Hb<7g/dl) and/or blood transfusion within the 12 month follow up period, and the mean fall in baseline Hb at day 7 and day 14. These outcomes will be compared between the intervention arms and also between each intervention arm and the controls.
Proportion of patients with Serious Adverse Drug reactions | 12 months
  The proportion of patients with one or more serious adverse drug reactions within 42 days of their primary treatment and also at 6 and 12 months.
Primaquine tolerability | 14 days
  Tolerability of primaquine will be assessed by comparing the proportion of patients with nausea, vomiting, abdominal pain and vomiting of a dose within 1 hour of administration between the intervention arms and also between each intervention arm and the controls.
Primaquine tolerability comparison between patients in intervention arm and control arm | 14 days
  Drug tolerability will be assessed also by comparing the proportion of patients completing a full course of observed primaquine therapy between the intervention arms and also between each intervention arm and the controls.
Incidence risk of severe anaemia in G6PD deficient arm | 14 days
  - The G6PD deficiency treatment arm will provide important data on the safety and tolerability of the WHO recommended weekly regimen. The incidence risk of severe anaemia (Hb<7g/dl) and/or requirement for blood transfusion within the 12 month follow up period and the mean fall in baseline Hb at day 7 and day 14 will be determined.
Cost effective analysis in the management of P. vivax with respect to the use of G6PD tests | 12 months
  The cost of illness will be compared between the intervention arms and also between each intervention arm and the controls. A cost-effectiveness analysis for the management of P. vivax with respect to the use of G6PD tests, the dosing schedule and the epidemiological context will be conducted.

CONTACTS AND LOCATIONS:
Overall Officials: Ric Price, FRCP, Principal Investigator — University of Oxford
Locations (8):
- Afghanistan (2):
  - Provincial Malaria & Leishmania control program (PMLCP) Nangarhar, Jalalabad, Nangarhar
  - Laghman Provincial Hospital, Laghmān
- Ethiopia (2):
  - Metahara Sugar Factory Hospital, Metehara, Oromiya
  - Arba Minch Hospital, Ārba Minch, Snnpr
- Indonesia (2):
  - Hanura Health Center, Bandar Lampung, Lampung
  - Tanjong Leidong District Health Center, Medan, North Sumatra
- Vietnam (2):
  - Dak O and Bu Gia Map Health Communes, Bình Phước, Binh Phuoc Province
  - Krong Pa Hospital, Krông Pa, Gia Lai

REFERENCES:
- [Background] Taylor WRJ, Thriemer K, von Seidlein L, Yuentrakul P, Assawariyathipat T, Assefa A, Auburn S, Chand K, Chau NH, Cheah PY, Dong LT, Dhorda M, Degaga TS, Devine A, Ekawati LL, Fahmi F, Hailu A, Hasanzai MA, Hien TT, Khu H, Ley B, Lubell Y, Marfurt J, Mohammad H, Moore KA, Naddim MN, Pasaribu AP, Pasaribu S, Promnarate C, Rahim AG, Sirithiranont P, Solomon H, Sudoyo H, Sutanto I, Thanh NV, Tuyet-Trinh NT, Waithira N, Woyessa A, Yamin FY, Dondorp A, Simpson JA, Baird JK, White NJ, Day NP, Price RN. Short-course primaquine for the radical cure of Plasmodium vivax malaria: a multicentre, randomised, placebo-controlled non-inferiority trial. Lancet. 2019 Sep 14;394(10202):929-938. doi: 10.1016/S0140-6736(19)31285-1. Epub 2019 Jul 18. PMID 31327563
- [Derived] Taylor WRJ, Meagher N, Ley B, Thriemer K, Bancone G, Satyagraha A, Assefa A, Chand K, Chau NH, Dhorda M, Degaga TS, Ekawati LL, Hailu A, Hasanzai MA, Naddim MN, Pasaribu AP, Rahim AG, Sutanto I, Thanh NV, Tuyet-Trinh NT, Waithira N, Woyessa A, Dondorp A, von Seidlein L, Simpson JA, White NJ, Baird JK, Day NP, Price RN. Weekly primaquine for radical cure of patients with Plasmodium vivax malaria and glucose-6-phosphate dehydrogenase deficiency. PLoS Negl Trop Dis. 2023 Sep 6;17(9):e0011522. doi: 10.1371/journal.pntd.0011522. eCollection 2023 Sep. PMID 37672548
- [Derived] Thriemer K, Commons RJ, Rajasekhar M, Degaga TS, Chand K, Chau NH, Assefa A, Naddim MN, Pasaribu AP, Rahim AG, Sutanto I, Hien TT, Hailu A, Hasanzai MA, Ekawati LL, Woyessa A, Teferi T, Waithira N, Taylor WRJ, Ley B, Dondorp A, Baird JK, White NJ, Day NP, Price RN, Simpson JA, von Seidlein L. The heterogeneity of symptom reporting across study sites: a secondary analysis of a randomised placebo-controlled multicentre antimalarial trial. BMC Med Res Methodol. 2023 Sep 4;23(1):198. doi: 10.1186/s12874-023-02022-3. PMID 37667204
- [Derived] IMPROV Study Group. Improving the radical cure of vivax malaria (IMPROV): a study protocol for a multicentre randomised, placebo-controlled comparison of short and long course primaquine regimens. BMC Infect Dis. 2015 Dec 7;15:558. doi: 10.1186/s12879-015-1276-2. PMID 26643116
- See also: Related Info — http://dx.doi.org/10.1016/S0140-6736(19)31285-1